CLINICAL TRIAL: NCT03265990
Title: Comparison Between Haemorrhoidectomy by Ligasure and Conventional Surgery
Brief Title: Haemorrhoidectomy by Ligasure and Conventional Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Refaay Ahmed, araahmed, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ligaHaemorrhoidectomy
Record Dates: First submitted 2017-08-19; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Ligature; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Conventional haemrrhoidectomy,Ferguson technique
  Interventions: Procedure: Conventional haemorrhoidectomy
- Group B (Experimental): Ligasure haemorrhoidectomy
  Interventions: Procedure: ligasure haemroidectomy

INTERVENTIONS:
Procedure: ligasure haemroidectomy — In ligasure group,After the haemorrhoids are prolapsed out from the anal canal with an artery forceps,Ligasure haemorrhoidectomy will be performed by applying the ligasure forceps close to the edge of each pile.Repeated applications of the device will be performed and excision will be continued into the anal canal,lifting the pile from the internal anal sphincter,to the level of the vascular pedicle,which will be finally divided.
  Arms: Group B
Procedure: Conventional haemorrhoidectomy — According to the Ferguson technique
  * Manual anal sphincter stretching up to 4 fingers
  * Delivery of hemorrhoidal masses with artery forceps,one being applied at the base of haemorrhoid,the other at the apex.
  * skin incision at the base of haemorrhoids and submucosal dissection to lift the haemorrhoid mass off the internal sphincter.
  After this the haemorrhoid pedicle will be transfixed and the mucosal edges of the defect will be opposed.
  Arms: Group A

SUMMARY:
Comparison between Haemorrhoidectomy by Ligasure and conventional surgery

DETAILED DESCRIPTION:
Hemorrhoids, a varicose condition are one of the commonest illnesses which causes per rectal bleeding . Hemorrhoidectomy is the standard operation for grades III and IV hemorrhoids; it is superior to any proposed conservative procedure. Conventional haemorrhoidectomy is the open surgical procedure in which the haemorrhoid pedicle is ligated by a transfixing suture which may lead to some postoperative complications mostly pain, bleeding and wound infection which ultimately cause prolonged stay in hospital.

A number of surgeons believe that by avoiding vascular pedicle ligation the chances of secondary bleeding can be decreased .This stimulated the researchers to develop new techniques with a less severe course and faster recovery . Recent advances in instrumental technology including the bipolar electrothermal device, ultrasonic scalpel, and circular stapler are gaining popularity as effective alternatives in hemorrhoidectomy . Of these instruments, the LigaSure vessel sealing system has been recently introduced as a tool conceived to upgrade the conventional treatment of haemorrhoids. This reduces anal spasm and allows performing a bloodless haemorrhoidectomy with reduced post- operative pain and fast healing . .Thus this operation can be recommended as the ideal technique. Many trials were performed to compare LigaSure hemorrhoidectomy with conventional hemorrhoidectomy, although an overall favorable trend exists toward LigaSure, conclusions are not univocal and definitive; this creates some uncertainty, also considering the increasing cost for this disposable device: thus it is essential to keep on experimenting to determine whenever an actual advantage exists.

ELIGIBILITY:
Inclusion Criteria:

* all patients with ages between 18 to 70 years with symptomatic grade III, or IV hemorrhoid who will be operated on at the Department of general Surgery, Assuit University Hospital

Exclusion Criteria:

* age older than 70 years
* patients with Grade I and II haemorrhoids
* patients on anticoagulants
* patients with liver cirrhosis
* patients with the hematological disorder
* patients with the concomitant anal disease
* patients had previous history of anorectal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 1 month
  pain will be evaluated with visual analogue scale

SECONDARY OUTCOMES:
Intra operative blood loss | 1 day
  Amount of blood loss by cc during surgery
Wound healing | 2 months
  the healing of mucosa and skin